CLINICAL TRIAL: NCT03496727
Title: Analgesic Effectiveness of Serratus Anterior Block for Video-assisted Thoracoscopic Surgery
Brief Title: Serratus Anterior Block for Video-assisted Thoracoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gözen Öksüz, Assistant Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: 2018/01-29
Record Dates: First submitted 2018-04-02; First posted 2018-04-12 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative
Keywords: pain, VATS
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Serratus anterior plane block: Anesthesia induction was performed to all patients. At the end of the operation, patients were performed SAPB under Ultrasound guidance by the same anesthetist.For 24 hours postoperatively, tramadol was administered with patient-controlled analgesia (PCA) All patients were extubated after the operation and transferred to ICU.
  Interventions: Procedure: Serratus anterior plane block
- Patient controlled analgesia: Anesthesia induction was performed on all patients.At the end of the operation, all patients were performed with patient-controlled analgesia (PCA) All patients were extubated after the operation and transferred to ICU.
  Interventions: Procedure: Patient controlled analgesia

INTERVENTIONS:
Procedure: Serratus anterior plane block — Serratus anterior plane block+patient controlled analgesia
  Groups: Serratus anterior plane block
Procedure: Patient controlled analgesia — Patient-controlled analgesia
  Groups: Patient controlled analgesia

SUMMARY:
Ultrasound-guided SAPB is a facial plane block which maintained analgesia with blockade of lateral branches of intercostal nerves at above or below serratus plane muscle. There are few cases and studies in the literature reporting successful analgesia provided by SAPB in VATS operations. The serratus plane block is used in our clinic for postoperative analgesia in VATS operations. The aim of this study was to evaluate the postoperative pain scores and use of analgesia in patients performed with the serratus plane block in VATS operations in a

1-year period.

DETAILED DESCRIPTION:
Approval for the study was granted by the Clinical Research Ethics Committee and all procedures were carried out in accordance with the Helsinki Declaration. A retrospective examination was made of the anesthesia forms of patients underwent VATS May 2016 and June 2017. Due to incomplete data of 1 of these 35 patients, that case was excluded from the study. The patients were divided into two groups. 24 patients were performed SAPB and iv PCA (intravenous patient controlled analgesia) and 10 patient's pain management were provided with only PCA. No block was administered to 10 patients because of anticoagulant therapy and patient refused block application. The demographic data of the patients (age, gender, operation type, and duration) were obtained from the anesthesia forms. The postoperative pain scores of the patients, evaluated with a visual analog scale (VAS) at 1, 6, 12 and 24 hours postoperatively and the postoperative doses of analgesia used were taken from the block pain follow-up forms

ELIGIBILITY:
Inclusion Criteria:

VATS( Video-assisted thoracoscopy) operation

a.Serratus anterior plane block b.patient controlled analgesia

Exclusion Criteria:

missing data written consent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: VATS ( Video-assisted thoracoscopy)
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesic consumption | up to 24 hour
  Postoperative analgesic consumption

SECONDARY OUTCOMES:
Post-operative pain scores | up to 24 hour
  The patient's level of pain in the postoperative period will be evaluated by the use of a 100mm Visual Analogue Scale (VAS) 1.,6.,12.,24. hour

OTHER OUTCOMES:
Complications | Postoperative 1 week
  Postoperative Complications

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kahramanmaras Sutcu Imam University Hospital, Kahramanmaraş
  - KahramanmarasSIU, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okmen K, Metin Okmen B. Evaluation of the effect of serratus anterior plane block for pain treatment after video-assisted thoracoscopic surgery. Anaesth Crit Care Pain Med. 2018 Aug;37(4):349-353. doi: 10.1016/j.accpm.2017.09.005. Epub 2017 Oct 12. PMID 29033355